CLINICAL TRIAL: NCT01186380
Title: Safety of the PET-512MC Transesophageal Transducer (TEE)
Brief Title: Safety of the PET-512MC Transesophageal Transducer
Acronym: TEE
Status: Completed | Type: Observational
Sponsor: Toshiba America Medical Systems, Inc. (Industry)
Responsible Party: Terry Schultz, Manager Regulatory Affairs, Toshiba America Medical Systems, Inc.
Other Study IDs: TEE-002
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Transesophageal Transducer
Keywords: TEE; Transesophageal; Transducer; Esophagus; Ease of passage and during transitioning into and down the esophagus to complete a normal TEE study

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- TEE Procedure: patients requiring TEE procedure by their physician
  Interventions: Device: PET-512MC

INTERVENTIONS:
Device: PET-512MC — Transesophageal Transducer
  Other Names: TEE Transducer; TEE Probe

SUMMARY:
The objective of this Study is to demonstrate the safety of the PET-512MC TEE transducer as it is inserted and transitioned into the esophagus through the mouth.

DETAILED DESCRIPTION:
The PET-512MC is a multiplane transesophageal transducer designed for use with Toshiba Diagnostic Ultrasound Systems for the visualization of the heart (and other organs) as a real-time ultrasound image. It is inserted into the esophagus through the mouth to visualize a plane of the heart through the esophageal wall.

The purpose of this Study is to demonstrate the safety of the PET-512MC TEE transducer and gather feedback from the investigators related to the insertion of the transducer. The data will be used to determine the usability of the transducer in the clinical environment.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients ages 18 and above who have been scheduled for a TEE procedure by their physician
* Informed consent understood and signed
* Compliance with post-treatment and follow-up protocol requirements

Exclusion Criteria

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female patients ages 18 and above
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory B Clarke, MD, Principal Investigator — Christ Hospital
Locations (1):
- The Christ Hospital, Cincinnati, Ohio, United States